CLINICAL TRIAL: NCT07267858
Title: Effect of a Clinical Pilates Programme on Individuals With Gold A COPD on Lung Function, Motor Performance, Chest Mobility, Sleep and Physical Activity, and Health-related Quality of Life: an Interactive Approach Between Rehabilitation Nursing and Sports Sciences.
Brief Title: Clinical Pilates Programme on People With COPD Gold A: a Rehabilitation Nursing Approach.
Acronym: COPD_CPilates
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Trás-os-Montes and Alto Douro (Other)
Collaborators: Unidade Local de Saúde do Alto Ave, EPE (Other)
Responsible Party: Principal Investigator, Cristiana Marques, Enfermeira Cristiana Marques, University of Trás-os-Montes and Alto Douro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 142/2024-CAF
Record Dates: First submitted 2025-11-16; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: COPD; Clinical Pilates; Rehabilitation Nursing
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Sample of participants, divided into an experimental group and a control group:
  1. Clinical Pilates Group (CPG), a group of people receiving follow-up rehabilitation nursing consultations and participating in the CP programme, which included 20 people.
  2. Control Group (CG), a group that only underwent follow-up rehabilitation nursing consultations, in which 18 people participated.
  Randomisation was performed by organising the individuals who met the inclusion criteria in alphabetical order and alternately removing them for each of the groups.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Pilates Group (CPG) (Experimental): Group of individuals with ongoing rehabilitation nursing consultations who participate in the CP programme consisting of 16 sessions of 60 minutes each.
  Interventions: Behavioral: Clinical Pilates for people with COPD Gold A.
- Control Group (CG) (No Intervention): Group that only underwent follow-up rehabilitation nursing consultations.

INTERVENTIONS:
Behavioral: Clinical Pilates for people with COPD Gold A. — 8-week programme with face-to-face sessions twice a week, lasting approximately 60 minutes per session, using equipment such as soft balls and elastic bands.
  Arms: Clinical Pilates Group (CPG)

SUMMARY:
The main objective of this study is to evaluate the effects of a Clinical Pilates-based exercise programme on chest mobility, lung function, motor performance, physical activity levels, sleep quality and Health-Related Quality of Life (HRQoL) in individuals with Gold A COPD. Based on our research question, 'What is the effect of a Clinical Pilates programme on thoracic mobility, pulmonary function, motor performance, physical activity levels, sleep quality, and HRQoL in people with Gold A COPD?', we propose the following research hypotheses:

H1: The Clinical Pilates programme contributed to improved thoracic mobility in people with Gold A COPD.

H2: The Clinical Pilates programme contributed to improved lung function in people with Gold A COPD.

H3: The Clinical Pilates programme positively influences the motor performance of people with Gold A COPD.

H4: The Clinical Pilates programme positively influences the physical activity levels of people with COPD Gold A.

H5: The Clinical Pilates programme positively influences the sleep quality of people with COPD Gold A.

H6: The Clinical Pilates programme contributes to improving the HRQoL levels of people with COPD Gold A.

ELIGIBILITY:
Inclusion Criteria:

* Anyone diagnosed with COPD at GOLD stage A, duly identified in SClínico, registered with the USF and residing in the geographical area covered by the Guimarães UCC, whose participation is validated by their family doctor. Inclusion in the study implies participation in at least 60% of the programme sessions, namely 10.

Exclusion Criteria:

* People with a history of exacerbation of the disease less than 4 weeks ago, as the guidelines of the European Respiratory Society and the American Thoracic Society (2017) make a conditional recommendation on pulmonary rehabilitation after exacerbation and recommend waiting at least 3 weeks, severe osteoarticular limitation that prevents physical exercise, psychiatric illness or severe cognitive dysfunction, unstable comorbidities such as unstable ischaemic disease or decompensated heart failure, and exercise-induced hypoxemia refractory to oxygen administration.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2026-07-24 (Estimated)

PRIMARY OUTCOMES:
Effect of a Clinical Pilates programme, as a tool in the field of Rehabilitation Nursing, on thoracic mobility in people with COPD Gold A. | Applied pre-intervention and post-intervention (with a 2-month interval). Both in Experimental and control group.
  Chirometric tests of the Thorax (Lanza et al., 2013).
  * The person stands with their hands on their hips, chest bare, with the investigator in front of them;
  * A tape measure is placed over the patient's rib cage in the axillary region;
  * The zero point of the tape measure is fixed in the anterior region of the chest at each level: axillary, with the tape passing through the axillary fold, and xiphoid, with the tape fixed to the xiphoid process. The other end of the tape goes around the chest and is pulled by the examiner over this fixed point, exerting as little pressure as possible on the person's body (the tape is adjusted but not tightened, ensuring that the contour of the soft tissues remains unchanged).
  * The person is asked to take a maximum breath in, followed by a maximum breath out, holding each for at least 2 seconds.
  * The measurement (cm) is recorded at the end of the breath out and the breath in.
  * The measurement is repeated.
Effect of a Clinical Pilates programme, as a tool in the field of Rehabilitation Nursing on pulmonary function in people with COPD Gold A. | Applied pre-intervention and post-intervention (with a 2-month interval). Both in Experimental and control group.
  Peak expiratory flow - Peak Flow (Miler et al., 2005).
  * The person sits with their neck in a neutral position, looking straight ahead;
  * They hold the Peak Flow meter and place it close to their mouth (ensuring that the indicator needle is set at 0);
  * The person takes a deep breath, places the Peak Flow in their mouth, between their teeth and with their tongue under the mouthpiece, and blows as hard as possible without pausing;
  * The highest value of at least three readings is recorded, with only readings that do not differ by more than 20L/min being considered;
  * Invalidate the result in case of excess saliva in the mouthpiece or coughing during exhalation;
  * The measurement range is between 50-800 L/min in accordance with the applicable standard ISO 23747:2015.
Effect of a Clinical Pilates programme, as a tool in the field of Rehabilitation Nursing on motor performance in people with COPD Gold A. | Applied pre-intervention and post-intervention (with a 2-month interval). Both in Experimental and control group.
  One-minute sit-to-stand test (Vaidya et al., 2016) and modified Borg scale (Borg, 1982).
  * The person sits on a chair leaning against the wall, with knees and hips bent at 90º, feet flat on the floor and hands resting on their legs;
  * The person is asked to stand up and sit down from the chair as quickly as possible without support for one minute.
  * The number of repetitions is counted.
  * At the end, the 'Modified Borg Scale' is applied.
  * The scale is placed in front of the person and they are asked to rate the degree of dyspnoea they perceive.
  * The rating ranges from 0 to 10, with 0 being 'No shortness of breath' and 10 being 'Maximum shortness of breath'.
  * The person indicates the number corresponding to the dyspnoea they feel.
Effect of a Clinical Pilates programme, as a tool in the field of Rehabilitation Nursing on physical activity levels in people with COPD Gold A. | Applied pre-intervention and post-intervention (with a 2-month interval). Both in Experimental and control group.
  Actigraph® GT3X+ accelerometer. The brand protocol requires wearing the device for a period of 4 days, including 2 days at the weekend.
  The device will be programmed for 6 hours on the first day of assessment and recordings will be made every 15 seconds.
  A record sheet will be provided to indicate the times when the accelerometer is put on and taken off.
  The device is placed on the non-dominant wrist and daily recording of at least 600 minutes (10 hours) is mandatory.
Effect of a Clinical Pilates programme, as a tool in the field of Rehabilitation Nursing on sleep quality in people with COPD Gold A. | Applied pre-intervention and post-intervention (with a 2-month interval). Both in Experimental and control group.
  The brand protocol requires wearing the device for a period of 4 days, including 2 days at the weekend.
  The device will be programmed for 6 hours on the first day of assessment and recordings will be made every 15 seconds.
  A record sheet will be provided to indicate the times when the accelerometer is put on and taken off.
  The device is placed on the non-dominant wrist and daily recording of at least 600 minutes (10 hours) is mandatory.
Effect of a Clinical Pilates programme, as a tool in the field of Rehabilitation Nursing on Health-related quality of life (HRQoL) in people with COPD Gold A. | Applied pre-intervention and post-intervention (with a 2-month interval). Both in Experimental and control group.
  EQ-5D-5L (Ferreira et al., 2023).
  Likert scale (1 to 5) self-assessment that considers 5 domains:
  * Mobility: from 'I have no mobility problems' to 'I am unable to walk';
  * Personal care: 'I have no problems washing or dressing myself' to 'I am unable to wash or dress myself';
  * Usual activities (e.g. domestic, leisure or family activities): 'I have no problem performing my usual activities' to 'I am unable to perform my usual activities';
  * Pain/Discomfort: 'I have no pain or discomfort' to 'I have extreme pain or discomfort';
  * Anxiety/Depression: 'I am not anxious and/or depressed' to 'I am extremely anxious and/or depressed';
  * Visual scale from 0 to 100, where 0 is 'worst health imaginable' and 100 is 'best health imaginable.' The person is asked to place an X on the scale to indicate how they feel about their health at the moment.

CONTACTS AND LOCATIONS:
Locations (1):
- Unidade de Cuidados na Comunidade de Guimarães, Guimarães, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR